CLINICAL TRIAL: NCT01375699
Title: Randomized Open-label Phase 1b Study of Doxorubicin-based Chemotherapy Regimens, With and Without Sildenafil, With Exploratory Analysis of Intermediate Cardiac Markers
Brief Title: Doxorubicin With or Without Sildenafil, With Analysis of Cardiac Markers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-13419; NCI-2011-0098 (Registry Identifier: CTRP)
Record Dates: First submitted 2011-06-15; First posted 2011-06-17 (Estimated); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Breast Cancer; Gastrointestinal Cancer; Genitourinary Cancer; Sarcoma; Gynecologic Cancer
Keywords: Breast cancer; Gastrointestinal cancer; Genitourinary cancer; Sarcoma; Gynecologic cancer
MeSH Terms: conditions — Breast Neoplasms; Gastrointestinal Neoplasms; Urogenital Neoplasms; Sarcoma | interventions — Doxorubicin; Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sildenafil + doxorubicin (Experimental): Patients receive sildenafil citrate PO QD* beginning at least 2 days prior to scheduled first dose of doxorubicin hydrochloride and continuing until 2 weeks after last scheduled dose of doxorubicin hydrochloride. Patients also receive doxorubicin hydrochloride IV as clinically indicated and as prescribed by treating provider.
  NOTE: *Patients receive sildenafil citrate PO TID on days that doxorubicin hydrochloride is also administered.
  Interventions: Drug: Doxorubicin; Drug: Sildenafil
- Doxorubicin-based chemotherapy (Active Comparator): Patients receive doxorubicin hydrochloride IV as clinically indicated and as prescribed by treating provider.
  Interventions: Drug: Doxorubicin

INTERVENTIONS:
Drug: Doxorubicin — As prescribed by treating provider.
  Other Names: 123127; Doxorubicin Hydrochloride; 3-Hydroxyacetyldaunorubicin Hydrochloride; Adriamycin Hydrochloride; ADM; Adriacin; Adriamycin
Drug: Sildenafil — Given PO, by mouth
  Other Names: Viagra; Revatio; Sildenafil Citrate; 171599-83-0
  Arms: Sildenafil + doxorubicin

SUMMARY:
Sildenafil increases the therapeutic effect of doxorubicin used as treatment for cancers of solid tumors through both an increase in anti-tumor effects and protection from cardiac toxicity.

DETAILED DESCRIPTION:
Definitive study of sildenafil enhancement of anthracycline anticancer effects and cardioprotection would require a randomized, placebo-controlled trial involving large numbers of patients and many years of follow-up. It is appropriate to demonstrate that concurrent administration of sildenafil and doxorubicin is safe and tolerable. Second, in definitive studies it might be helpful to incorporate early markers of cardiac injury in order to gain early insight into cardioprotective effects, but there are no such established markers. As a correlative study, multiple intermediate markers will be tested. In order to investigate these candidate markers it is appropriate to study patients receiving doxorubicin alone, as early markers of injury may not be apparent in patients treated with the combination. In order to accomplish these two goals the trial is a randomized trial involving a sildenafil/doxorubicin group and a doxorubicin group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with any malignancy that is deemed appropriate for treatment with a chemotherapy regimen incorporating a < 3-hour infusion of doxorubicin >= 40 mg/m^2/dose not more frequently than weekly; single agent doxorubicin and combination chemotherapy are allowed; the duration of treatment and the cumulative dose of doxorubicin are determined by the chemotherapy regimen chosen for treatment of each individual's disease and up to the discretion of the treating provider; prior doxorubicin-based regimen(s) allowed, unless the most recent prior doxorubicin-based regimen resulted in documented refractory disease
* At least 30 days since last doxorubicin before initiation of current doxorubicin-based regimen
* Performance status Eastern Cooperative Oncology Group (ECOG) equal to or less than 2
* Life-expectancy > 1 year
* Women of childbearing potential and men must agree to use a medically accepted form of birth control for the duration of study and for a minimum of 6 months after the last dose of doxorubicin
* Ability to understand and the willingness to sign a written informed consent; a signed informed consent must be obtained prior to any study-specific procedures

Exclusion Criteria:

* Known congestive heart failure (CHF) (active disease or history of)
* Left ventricular ejection fraction less than 55%
* Planned concurrent administration of other investigational agents
* Planned subsequent therapy with a human epidermal growth factor receptor 2 (HER2)-directed treatments (trastuzumab, pertuzumab, trastuzumab emtansine [T-DM1]) or other anthracyclines besides doxorubicin
* Swallowing or absorption problems that might interfere with oral bioavailability of sildenafil
* Known hypersensitivity to doxorubicin, sildenafil or any component of either agent
* Planned chronic nitrate or alpha blocker therapy
* Exclude persons who require ongoing administration of STRONG cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) inhibitors and/or inducers; short periods of exposure to CYP3A4 inhibitors will be allowed (i.e., exposure to aprepitant for three days at the time of doxorubicin exposure)
* Other relative contraindications to sildenafil as defined in the prescribing information:

  * Myocardial infarction, stroke, or life-threatening arrhythmia within the last 6 months
  * Coronary artery disease causing unstable angina
  * Resting hypotension (blood pressure [BP] < 90/50) or hypertension (BP > 170/110) despite appropriate treatment
  * Known retinitis pigmentosa
* Persisting or anticipated toxicity from prior therapy that might confound attribution of on-study adverse events (AEs)
* Pregnant or nursing
* Known hearing loss
* History of priapism when exposed to PDE5 inhibitors (sildenafil, vardenafil, tadalafil)
* Other condition(s) that in the opinion of the investigator might compromise the objectives of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-08-11 (Actual); Primary Completion 2017-08-04 (Actual); Study Completion 2018-01-19 (Actual)

PRIMARY OUTCOMES:
Safety of concurrent sildenafil with doxorubicin-based chemotherapy | 25 months
  Sildenafil will be administered at least 7 days prior to scheduled first dose of doxorubicin and continue daily dosing through 2 weeks after last doxorubicin dose. Multiple biomarkers as candidate early markers of anthracycline-induced cardiotoxicity will be tested.
The difference in left ventricular ejection fraction (LVEF) between arms | 4 years
  A repeated measures analysis of variance (ANOVA) will be used to compare the LVEF between Arm 1 and Arm 2 over all visits. A pooled t-test will also be performed to determine the change in LVEF between first and last visits.

SECONDARY OUTCOMES:
Comparison of candidate early markers of cardiac injury | 37 months
  The fluctuation in the levels of biomarkers including novel ultra sensitive troponins and BNP, as well as tissue doppler imaging studies with echocardiography will analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew S. Poklepovic, MD, Principal Investigator — Massey Cancer Center
Locations (1):
- Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia, United States

REFERENCES:
- [Result] Poklepovic A, Qu Y, Dickinson M, Kontos MC, Kmieciak M, Schultz E, Bandopadhyay D, Deng X, Kukreja RC. Randomized study of doxorubicin-based chemotherapy regimens, with and without sildenafil, with analysis of intermediate cardiac markers. Cardiooncology. 2018;4:7. doi: 10.1186/s40959-018-0033-2. Epub 2018 Aug 29. PMID 30221011